CLINICAL TRIAL: NCT07119567
Title: Longitudinal Exploration of Subjective and Objective Sleep Characteristics in Patients With Cocaine Use Disorder During the Withdrawal Process
Brief Title: Impact of Cocaine Use and Withdrawal on Sleep
Acronym: CokeSo
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A00292-47
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine use disorder; Withdrawal; Sleep; Polysomnography; Actimetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cocaine Use Disorder Group: A cohort of 32 patients with cocaine use disorder will undergo repeated sleep assessment at three key stages: during active use, at the beginning of withdrawal, and after a period of sustained withdrawal. All participants will serve as their own control across timepoints
  Interventions: Other: Multimodal Sleep and Biomarker Assessment

INTERVENTIONS:
Other: Multimodal Sleep and Biomarker Assessment — Participants will undergo non-invasive sleep assessments including polysomnography recordings (using the Somfit® device), actigraphy, self-reported questionnaires (on sleep, substance use), and urinary biomarker collection (for cortisol and melatonin levels) at three distinct stages of their substance use/withdrawal timeline.

SUMMARY:
This study investigates how cocaine use and withdrawal affect sleep and circadian rhythms in individuals undergoing inpatient detoxification. Using wearable sleep monitors, actigraphy, questionnaires, and hormonal biomarkers, it aims to capture both objective and subjective changes in sleep across three key stages: active use, early withdrawal, and late withdrawal. The study is unique in its ability to explore sleep microstructure, the circadian system's role via melatonin and cortisol measurements, and the dynamic relationship between subjective sleep perception and objective sleep data. It also examines whether sleep quality may serve as a predictive marker of long-term withdrawal success.

DETAILED DESCRIPTION:
Sleep disturbances are a common but poorly understood feature of cocaine use disorder, and may play a critical role in both relapse vulnerability and treatment outcomes. This interventional study aims to explore objective and subjective sleep patterns, as well as circadian regulation, across three distinct phases: during active cocaine use, early withdrawal, and late withdrawal. Participants will be individuals scheduled for supervised inpatient detoxification.

The study employs a multimodal assessment strategy:

* Ambulatory polysomnography using the Somfit® device will allow analysis of both macro- and microstructure of sleep across two nights per visit.
* Actigraphy will be used to capture precise temporal dynamics of sleep-wake rhythm over the course of the study.
* Subjective measures will include validated self-report questionnaires on sleep quality, insomnia severity, sleepiness, fatigue, and sleep perception.
* Urinary biomarkers (free cortisol and 6-sulfatoxymelatonin, collected 5 times/day) will provide data on circadian rhythm integrity, enabling exploration of the role of circadian dysregulation in sleep disturbances.

A key originality of the study lies in its ability to dynamically assess the relationship between subjective and objective sleep parameters and to explore the circadian contribution to sleep disruption in cocaine users. Furthermore, by following patients through early and late withdrawal, the study will investigate whether sleep parameters could serve as predictive markers of long-term withdrawal success, offering potential targets for future therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or older
* Meeting DSM-5 criteria for cocaine use disorder
* Positive urine drug screen for cocaine
* Scheduled for inpatient supervised cocaine detoxification within the next four weeks
* Covered by a national health insurance plan or social security system
* Have a valid, personal means of contact (telephone or email address) enabling remote follow-up at 6 months.

Exclusion Criteria:

* Current diagnosis of opioid use disorder or other psychostimulant use disorders (e.g., amphetamines, methamphetamines, cathinones, methylphenidate)
* Unstable psychiatric disorder or somatic illness deemed incompatible with study participation by the investigator
* Current treatment with methylphenidate, modafinil, solriamfetol, melatonin, pitolisant, naltrexone, or bupropion
* Patients under legal guardianship
* Pregnant or breastfeeding women: a pregnancy test will be performed prior to inclusion for women of childbearing potential
* Individuals deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cocaine use disorder seeking hospitalization for withdrawal
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency (%) measured by polysomnography | 30 months
  Sleep efficiency, defined as the ratio of total sleep time to time spent in bed, will be assessed using the Somfit® wearable device. Measurements will be conducted over three visits corresponding to distinct stages of cocaine use and withdrawal: V1 (active use), V2 (early withdrawal), and V3 (late withdrawal). Each visit includes two consecutive nights of recording, and the 2 nights will be averaged for analysis purposes. This double recording also makes it possible to obtain data from one night if the second encounters a technical problem. The primary outcome will be derived from data collected over a 16-hour window encompassing the nocturnal sleep period.

SECONDARY OUTCOMES:
Objective Sleep Parameters measured by polysomnography | 30 months
  Objective sleep metrics including total sleep time (min), sleep onset latency (min), wake after sleep onset (WASO, min), REM sleep duration and latency, time spent in N1, N2, N3 stages (min and %), micro-arousal index, phasic/tonic REM proportions, spindle index in NREM sleep, and delta power during N3 will be recorded via polysomnography (SOMFIT) across three study visits (each comprising two nights of measurement).
Sleep-Wake Rhythm Parameters from Actigraphy | 30 months
  Actigraphy data from the MotionWatch 8® will be used to assess weekly sleep-wake patterns. Extracted parameters include sleep onset and offset times, sleep midpoint, time in bed, total sleep time, sleep onset latency, WASO, sleep efficiency, and diurnal naps (presence, number, duration, and timing).
Sleep-Wake Rhythm Parameters from Sleep Diary | 30 months
  Entries in the sleep diary will be used to assess weekly sleep-wake patterns
Subjective Sleep Scores | 30 months
  Sleep-related self-reported outcomes will be assessed using the following validated questionnaires completed after polysomnography nights.
Circadian Rhythmicity via Urinary Cortisol | 30 months
  Circadian rhythm will be evaluated by analyzing sequential urinary samples (5/24h) for free cortisol levels at two withdrawal phases: early withdrawal (Visit 2) and late withdrawal (Visit 3).
Circadian Rhythmicity via Melatonin Metabolites | 30 months
  Circadian rhythm will be evaluated by analyzing sequential urinary samples (5/24h) for 6-sulfatoxymelatonin levels at two withdrawal phases: early withdrawal (Visit 2) and late withdrawal (Visit 3).

CONTACTS AND LOCATIONS:
Overall Officials: BENJAMIN ROLLAND, MD, PhD, Principal Investigator — Centre Hospitalier le Vinatier